CLINICAL TRIAL: NCT04640363
Title: Combi-elastography Assessment of HCC Recurrence After Thermal Ablation Multi-center Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Chinese PLA General Hospital
Other Study IDs: S2020-387-03
Record Dates: First submitted 2020-11-10; First posted 2020-11-23 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: HCC; Recurrence Tumor
Keywords: Thermal ablation; Elastography; Ultrasound; Recurrence; Predictive Cancer Model
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Combined F index, A index,ATT index and spleen stiffness to predict tumor recurrence in different liver settings after thermal ablation of HCC.

DETAILED DESCRIPTION:
Thermal ablation is one of the established method for HCC treatment. Postoperative recurrence of HCC is one of the major factors leading to poor prognosis of HCC patients. Most studies have shown that the risk factors of recurrence include tumor size, tumor number and intrahepatic spread, etc.

Besides, the carcinogenic effects of inflammatory activity and fibrosis in liver background caused by chronic hepatitis also be related to the recurrence. In the study, combi-elastography imaging technology , not only the F index which is related to liver fibrosis stage can be obtained, but also the A index which is related to inflammation activity can be measured, this may provide a more valuable method for tumor recurrence of early prediction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years of age, and gender not limited;Chronic hepatitis B patients;The lesions of liver have the histopathological diagnosis of HCC and within MiLan criteria;All lesions were performed thermal ablation surgery;Sign the informed consent.

Exclusion Criteria:

* Lesions that unrealized complete inactivation evaluation by the enhanced imaging;Merging other systems' serious illness that can't cooperate with elastic imaging checking(such as heart failure, renal failure, such as mental illness);After liver transplantation patients;Patients with pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent thermal ablation of HCC will be observed and evaluate the predictive power of combined elastography for tumor recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
F index | baseline
  F index is linked to the degree of liver fibrosis,and it can be available by ultrasound elastography checking.
A index | baseline
  A index is linked to the degree of hepatitis,and it can be available by ultrasound elastography checking.
ATT index | baseline
  ATT index is linked to the degree of steatosis of liver,and it can be available by ultrasound elastography checking.
Spleen stiffness | baseline
  Spleen stiffness can be available by ultrasound elastography checking.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China